CLINICAL TRIAL: NCT00381875
Title: A Pilot Study to Investigate the Safety and Immunogenicity of a Peptide Vaccine for HIV Infected HLA-A2 Individuals Designed to Impede the Development of Antiretroviral Resistance
Brief Title: Vaccine Therapy, Incomplete Freund's Adjuvant, and GM-CSF in Treating Patients With HIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 060211; 06-C-0211; NCI-P6066; NCI-6958; CDR0000495768
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Nonneoplastic Condition
Keywords: HIV infection
MeSH Terms: conditions — HIV Infections | interventions — incomplete Freund's adjuvant; sargramostim; Immunoenzyme Techniques

INTERVENTIONS:
Biological: E1M184V peptide vaccine
Biological: incomplete Freund's adjuvant
Biological: sargramostim
Other: immunoenzyme technique

SUMMARY:
RATIONALE: Vaccines made from peptides may help the body build an effective immune response. Incomplete Freund's adjuvant may stimulate the immune system in different ways and may help the vaccine work better. Colony-stimulating factors, such as GM-CSF, may increase the number of immune cells found in bone marrow or peripheral blood. Giving vaccine therapy together with incomplete Freund's adjuvant and GM-CSF may be an effective treatment for patients with HIV.

PURPOSE: This clinical trial is studying how well giving vaccine therapy together with incomplete Freund's adjuvant and GM-CSF works in treating patients with HIV.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the safety of vaccination comprising E1M184V peptide with incomplete Freund's adjuvant in combination with sargramostim (GM-CSF) in patients with HIV who are HLA-A2 positive.
* Assess, preliminarily, the ability of E1M184V peptide vaccine to induce a cytotoxic T-cell response, defined by ELISPOT assay, in these patients.

Secondary

* Explore, preliminarily, the effect of this regimen on HIV viral load and CD4 count in these patients.
* Explore, preliminarily, the development of lamivudine or emtricitabine resistance in patients who subsequently receive lamivudine or emtricitabine.
* Explore, preliminarily, the ability of E1M184V peptide vaccine to induce a cytotoxic T-cell response as assessed by HLA-A2 class I tetramers and intracellular interferon gamma production after stimulation with E1M184V.

OUTLINE: This is a pilot study.

Patients receive vaccination comprising E1M184V peptide and incomplete Freund's adjuvant subcutaneously (SC) on day 1 in weeks 0, 4, 8, 12, and 16. Patients also receive sargramostim (GM-CSF) SC immediately after vaccination and once daily on days 1-4. Some patients do not receive GM-CSF after the first 2 doses of vaccine. Treatment continues in the absence of unacceptable toxicity.

Patients undergo blood collection at baseline and at 4, 12, 20, 36, and 52 weeks for biomarker/laboratory analysis. Assays may include immunoenzyme techniques and viral genotyping.

After completion of study treatment, patients are followed periodically for up to 2 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* HIV-1 infection confirmed by Western blot and enzyme-linked immunosorbent assay
* HLA-A2 positive by polymerase chain reaction-sequence specific primers
* CD4 T-cell count ≥ 300/mm³
* Must be receiving stable regimen of highly active antiretroviral therapy (HAART) that does not include lamivudine or emtricitabine for ≥ 1 month prior to study entry

  * Patients on HAART, including lamivudine or emtricitabine, for which there is a medically appropriate regimen that does not include lamivudine or emtricitabine, are eligible if willing to change antiretrovirals
* Viral load < 50 copies/mL for 1 month prior to study entry

PATIENT CHARACTERISTICS:

* See Disease Characteristics
* ECOG performance status 0-1
* Life expectancy ≥ 6 months
* Hemoglobin ≥ 9 g/dL
* WBC ≥ 1,000/mm³
* Absolute neutrophil count ≥ 750/mm³
* Platelet count ≥ 75,000/mm³
* PT and PTT ≤ 120% of control unless lupus anticoagulant detected
* Bilirubin ≤ 1.5 times upper limit of normal (ULN) (≤ 7.5 mg/dL with direct fraction ≤ 0.7 mg/dL if on protease inhibitor therapy or due to Gilbert's syndrome)
* AST and ALT ≤ 2.5 times ULN
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No hepatitis B surface antigen (HBsAg) or a prior history of HBsAg while on lamivudine or emtricitabine

  * Prior treatment with tenofovir and currently HBsAg negative allowed
* No evidence of a severe or life-threatening infection other than HIV within the past 6 months
* No opportunistic infections requiring systemic therapy within the past month
* No active malignancy, except for basal cell carcinoma
* No known hypersensitivity to incomplete Freund's adjuvant or incomplete Freund's adjuvant VG (vegetable-grade), E1M184V peptide, or sargramostim (GM-CSF)
* No other abnormality that would be scored as ≥ grade 3 toxicity, except any of the following (if asymptomatic):

  * Hyperuricemia of grade 4 (without physiologic consequences)
  * Elevation of lactate dehydrogenase ≥ grade 3
  * Elevation of creatine phosphokinase (CPK) ≥ grade 3
  * Hypophosphatemia ≥ grade 3 (if patient is on tenofovir)
  * Elevation of alkaline phosphate of grade 3
  * Hyperamylasemia of ≥ grade 3 allowed if any of the following criteria are met:

    * Macroamylasemia
    * Lipase ≤ 2 times ULN
  * Lymphopenia grade 3
* No other condition that, in the opinion of the investigator, would preclude compliance with study requirements

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No systemic corticosteroids within the past 3 weeks

  * Concurrent systemic corticosteroids allowed in the short term only
  * Physiologic replacement doses of steroids allowed
* No prior vaccination with a vaccine that includes all or part of the reverse transcriptase of HIV-1
* No other concurrent investigational drugs or vaccinations
* No concurrent lamivudine or emtricitabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Impact of treatment on immune response, in terms of the difference between cytotoxic T-lymphocyte effector frequency, as measured by enzyme-linked immunospot (ELISPOT) at baseline and at week 20

SECONDARY OUTCOMES:
Effects of treatment on viral load
Sequencing of any resultant HIV strains
CD4 counts for assessment of effects on HIV disease

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M. Wyvill, BSN, RN — NCI - HIV and AIDS Malignancy Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States